CLINICAL TRIAL: NCT02821741
Title: Effects of External Ear Stimulation on Pain Perception and Mood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 160136; 16-AT-0136
Record Dates: First submitted 2016-06-29; First posted 2016-07-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Pain in Healthy Participants
Keywords: Sensory Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cymba Conchae (Experimental): Mild electrical stimulation is applied to the cymba conchae of the left ear, and thermal stimulation is applied to the arms.
  Interventions: Device: The Twin Stim Plus, 3rd Edition; Device: Medoc Pathway System
- Ear Lobe (Active Comparator): Mild electrical stimulation is applied to the earlobe of the left ear, and thermal stimulation is applied to the arms.
  Interventions: Device: The Twin Stim Plus, 3rd Edition; Device: Medoc Pathway System

INTERVENTIONS:
Device: The Twin Stim Plus, 3rd Edition — Mild transcutaneous electrical stimulation will be applied to the cymba conchae of the left ear on day 1 and the left earlobe on day 2 (or vice versa) using a commercially available TENS unit (transcutaneous electrical nerve stimulator) attached to a pair of silver electrodes.
Device: Medoc Pathway System — Device used to apply Thermal stimulation to both arms.

SUMMARY:
Background:

The vagus nerve runs from the brain to many organs. Stimulating it can affect the experience of pain. The nerve can be stimulated on the surface of the left ear. Researchers want to study how this stimulation affects the perception of pain. They also want to study how mood affects the experience of pain.

Objective:

To study the effects of mood and vagus nerve stimulation on the experience of pain.

Eligibility:

Healthy people ages 18 and older who are fluent in English

Design:

Participants will be pre-screened with a 15-minute phone call.

Participants will have three 2-hour visits.

At the screening visit, participants will be screened with:

Medical and psychiatric history

Physical and psychological exams

Questionnaires about physical and psychiatric health and mood

Urine tests

A heat probe on the forearm. The temperature will be increased until it is painful

but tolerable.

Participants will have 2 testing sessions within 7 days. Before the testing, they cannot do the following:

Eat, use nicotine, or exercise for at least 2 hours

Drink alcohol for 24 hours

Take certain medicines for 3 days

Testing includes:

Urine drug screening

Left ear stimulation: In one session, the vagus nerve will be stimulated. In the other, an area

of the ear away from the vagus nerve will be stimulated. This will be done with mild electric

shocks that cause a tingling, pricking, or itchy feeling.

Heat applied to the forearm until it is painful but tolerable

Completing several forms on a computer or on paper about how they are feeling

Monitors on the chest and a finger clip to monitor heart, breathing, and blood pressure

DETAILED DESCRIPTION:
This double-blind, randomized, controlled, cross-over study on healthy participants will evaluate the perceptual differences of pain and changes in mood in response to peripheral nerve stimulation over two regions of the left external ear. A series of short and long duration heat stimuli will be applied to the participants forearms and they will be asked to rate their current mood state, the intensity of the pain, and whether it was pleasant or unpleasant. The series of heat stimuli will be applied before, during, and after mild electrical stimulation of the left external ear using a commercially available TENS unit. There are two study sessions. Session 1 involves eligibility screening, a brief practice session, followed by the testing session. In Session 2 (no more than 7 days later), the testing session will be repeated with the exception of the location of ear stimulation. Up to 76 people, ages 18-50 years old, will be enrolled in the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be:

1. between 18 and 50 years old.
2. fluent in English.
3. able to provide written informed consent.

EXCLUSION CRITERIA:

Overall exclusion criteria for the study

1. Unable to comply with study procedures or visits (including inability to schedule the second session within 10 business days of the first session).
2. Is pregnant or breastfeeding.
3. Has ears with indiscernible structures (e.g., cymba conchae, earlobe) due to congenital malformations, accidents, or physical alterations (e.g., "gauge", cartilage piercing).
4. Has a dermatological condition such as scars or burns, or has had a tattoo in the testing region within the previous four weeks that might influence cutaneous sensibility.
5. Women who consume more than 7 alcoholic beverages per week, and men who consume more than 14 drinks per week.
6. Has a current chronic pain condition or has had chronic pain in the past year (painful condition lasting more than six months).
7. Has a major medical condition, such as kidney, liver, cardiovascular, autonomic, pulmonary, or neurological problems (e.g., epilepsy) or a chronic systemic disease (e.g., diabetes).
8. Has or had psychiatric disorders such as major depression, major anxiety-related problems, post-traumatic stress syndrome, bipolar disorder, psychosis, or alcohol or substance abuse disorders as identified by the MINI International Neuropsychiatric Interview questionnaire, which will be administered as part of the screening procedure.
9. Has a medical condition potentially affecting cardiac functioning (e.g. arrhythmias, bradycardia [<60 beats per min; determined during screening]) or Raynaud s Disease or other medical condition affecting peripheral vascular sensitivity.
10. Is actively taking medications that are known to interfere with current measurements of pain or autonomic function. These include but are not limited to: opioids, antidepressants (such as tricyclic antidepressants, selective serotonin reuptake inhibitors, and serotonin norepinephrine reuptake inhibitors), anticonvulsants (including gabapentin and pregabalin), and blood pressure medications (including beta-blockers, calcium channel blockers, and ACE inhibitors). Participants who have used such medications in the last three months must have ceased taking them for at least one month or three medication half-lives (whichever is longer) in order to be included.
11. Baseline heat pain threshold exceeds 46 degrees C (to be determined after consent).
12. Has ever had acupuncture in or around any area of the ears.
13. NIH employees are subordinates, relatives, or co-workers of the investigators, or NCCIH DIR employees.

Exclusion criteria for individual study session*

1. Has consumed alcohol within 24 hours, shows signs of alcohol withdrawal syndrome, or has behavioral signs of intoxication.
2. Has exercised or eaten within two hours of testing session.
3. Used nicotinic substances (e.g., tobacco, gum, "e-cigarette") within 2 hours of testing.
4. Used topical pain-relieving creams in the testing area (e.g. methylsalicylate, capsaicin) within 24 hours of testing.
5. Used non-steroidal anti-inflammatory drugs (NSAIDS, e.g. aspirin, ibuprofen), acetaminophen, naproxen, sumatriptan within 3 days of testing.

   * To be determined during the pre-session screening. Participants that cannot refrain from these activities may have their session rescheduled up to two times. If the participant is found non-compliant during the second rescheduled appointment, he or she will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-10-18 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The difference in pain ratings collected for each subject during the two types of left ear stimulation (cymba conchae and earlobe). | End of study
  See measures

SECONDARY OUTCOMES:
The effect of tVNS on pain threshold, pain unpleasantness, and mood as measured by visual analogue scales (VAS). | End of Study
  See measures
Mood and anxiety, as measured by questionnaires taken at the beginning and end of both study sessions. | End of study
  See measures
Autonomic measures will be analyzed to determine whether tVNS has an effect on heart rate variability. | End of study
  See measures

CONTACTS AND LOCATIONS:
Overall Officials: Alisa J Johnson, Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-AT-0136.html